CLINICAL TRIAL: NCT05369767
Title: A Phase 1, Randomized, Double Blind, Dose-escalation, Placebo Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-2004 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of Single-dose Injection of SHR-2004 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SHR-2004-101
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Prevention of Arterial and Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Sagittal Abdominal Diameter

STUDY DESIGN:
Intervention Model Description: SHR-2004 injection compared with placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAD, SHR-2004 (Experimental): Up to 6 cohorts of healthy subjects will receive a single dose of SHR-2004 injection
  Interventions: Drug: SAD, SHR-2004
- SAD, SHR-2004 placebo (Placebo Comparator): Up to 6 cohorts of healthy subjects will receive a single dose of SHR-2004 placebo injection
  Interventions: Drug: SAD, SHR-2004 placebo

INTERVENTIONS:
Drug: SAD, SHR-2004 — Ascending dose
  Arms: SAD, SHR-2004
Drug: SAD, SHR-2004 placebo — Ascending dose
  Arms: SAD, SHR-2004 placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of SHR-2004 injection in healthy subjects. In addition, this study will provide information on pharmacokinetics and pharmacodynamics of SHR-2004 injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. males or females, aged 18-55;
2. body mass index (BMI) between 19 kg/m2 to 28 kg/m2, and a total body weight: male ≥50.0 kg and <90.0 kg; female ≥45.0 kg and <90.0 kg.

Exclusion Criteria:

1. previous medical history of coagulation or bleeding disorders;
2. known risks of bleeding or thrombosis, such as recurrent gingival bleeding, spontaneous bleeding, haemorrhoids, gastrointestinal ulcers, or other high-risk bleeding diseases.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
To assess the number of subjects with adverse events (AEs) and serious adverse events (SAEs) | up to day 113

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Drum Tower Hospital of Nanjing University Medical school, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma T, Weng Z, Cao B, Dong Y, Deng C, Huang L, Yang Y, Wang Y, Shen C, Wang L, Shen K, Li J. The first-in-human study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of the factor XI monoclonal antibody SHR-2004 in healthy subjects. Expert Opin Investig Drugs. 2024 Oct;33(10):1075-1082. doi: 10.1080/13543784.2024.2391837. Epub 2024 Aug 22. PMID 39166425